CLINICAL TRIAL: NCT03892720
Title: A Phase II Study of Non-Coplanar SBRT Re-Irradiation Using HyperArc in Patients With Recurrent Head and Neck Cancer
Brief Title: Stereotactic Body Radiation Therapy Using HyperArc in Treating Patients With Recurrent Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-001247; NCI-2018-02996 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Head and Neck Carcinoma
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (SBRT) (Experimental): Patients undergo stereotactic body radiation therapy with either standard radiation treatment software or HyperArc software technology for 2-3 fractions per week over a 2-week period for 5 fractions.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase II trial studies how well stereotactic body radiation therapy with HyperArc software technology works in treating patients with head and neck cancer that has come back. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate local control and toxicity of patients who receive escalated dose stereotactic body radiation therapy (SBRT) reirradiation with HyperArc for recurrent head and neck cancer (rHNC).

SECONDARY OBJECTIVES:

I. To evaluate the clinical benefit of HyperArc through the analysis of overall survival (OS), progression-free survival (PFS) and locoregional progression-free survival (LPFS).

EXPLORATORY OBJECTIVES:

I. To evaluate dosimetric data including dose to target and organs at risk (OAR).

OUTLINE:

Patients undergo treatment planning with both standard radiation treatment software and HyperArc software technology. The most optimal plan will be delivered to a total dose of 55 Gy in 5 fractions, given 2-3 times weekly.

After completion of study treatment, patients are followed up periodically for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent head and neck cancer; either unresectable or status post salvage surgery.
* History of radiation therapy for head and neck cancer with minimum 50% overlap of the 50% isodose line from prior treatment to the proposed treatment volume.
* Estimated life expectancy > 12 weeks.
* Karnofsky performance status >= 70 (Eastern Cooperative Oncology Group [ECOG] 0-2).
* Maximum tumor, or tumor bed, diameter < 5 cm.
* If a woman is of childbearing potential, a negative serum pregnancy test must be documented. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) for duration of study participation and for up to 4 weeks following the study treatment.
* Ability to understand and willingness to sign a written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Local control rate of the treated tumor target per Response Evaluation Criteria in Solid Tumors version 1.1, magnetic resonance imaging (MRI) response or positron emission tomography (PET) response | At 1 year
  Will calculate the percentage and construct 95% exact confidence interval for local control rate.
Percent of patients with acute or chronic grade >= 3 treatment-related toxicity per Common Terminology Criteria for Adverse Events version 4.0 | At 1 year
  Data will be tabulated and summarized. Incidence of adverse events (AEs) will be summarized overall and with separate summaries for serious adverse events (SAEs), AEs leading to discontinuation, AEs leading to death, etc. The overall safety and tolerability will be assessed throughout the study period. All AE data will be listed individually by patient identifier.

SECONDARY OUTCOMES:
Overall survival (OS) | The time between the first dose of stereotactic body radiation therapy (SBRT) and death, assessed at 1 year
  The Kaplan-Meier method will be used to provide an estimate of OS. The corresponding 95% confidence interval will also be presented.
OS | The time between the first dose of SBRT and death, assessed at 2 years
  The Kaplan-Meier method will be used to provide an estimate of OS. The corresponding 95% confidence interval will also be presented.
Median OS | The time between the first dose of SBRT and death, assessed up to 2 years
  The Kaplan-Meier method will be used to provide an estimate of median OS. The corresponding 95% confidence interval will also be presented.
Progression-free survival (PFS) | From the first dose of SBRT to the first objectively documented disease progression or death due to any cause, assessed at 1 year
  The Kaplan-Meier method will be used to provide an estimate of PFS. The corresponding 95% confidence interval will also be presented.
PFS | From the first dose of SBRT to the first objectively documented disease progression or death due to any cause, assessed at 2 years
  The Kaplan-Meier method will be used to provide an estimate of PFS. The corresponding 95% confidence interval will also be presented.
Median PFS | From the first dose of SBRT to the first objectively documented disease progression or death due to any cause, assessed up to 2 years
  The Kaplan-Meier method will be used to provide an estimate of median PFS. The corresponding 95% confidence interval will also be presented.
Locoregional progression-free survival (LPFS) | From the first dose of SBRT to the first objectively documented disease progression in either the primary tumor, adjacent to the primary tumor, or in the surrounding lymph node areas, assessed at 1 year
  The Kaplan-Meier method will be used to provide an estimate of LPFS. The corresponding 95% confidence interval will also be presented.
LPFS | From the first dose of SBRT to the first objectively documented disease progression in either the primary tumor, adjacent to the primary tumor, or in the surrounding lymph node areas, assessed at 2 years
  The Kaplan-Meier method will be used to provide an estimate of LPFS. The corresponding 95% confidence interval will also be presented.
Median LPFS | From the first dose of SBRT to the first objectively documented disease progression in either the primary tumor, adjacent to the primary tumor, or in the surrounding lymph node areas, assessed up to 2 years
  The Kaplan-Meier method will be used to provide an estimate of median LPFS. The corresponding 95% confidence interval will also be presented.

OTHER OUTCOMES:
Dosimetric data including achievable dose to target and organs at risk (OAR) | Up to 2 years
  Data will be collected but not analyzed.
Serum markers predictive of response and/or toxicity | Up to 2 years
  Will perform correlation analysis to explore serum markers predictive of efficacy endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chin, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States